CLINICAL TRIAL: NCT02600676
Title: Randomized, Double Blind, Placebo Controlled Trial of Sacral Transcutaneous Electric Nerve Stimulation (TENS) in Children With Enuresis
Brief Title: Transcutaneous Electric Nerve Stimulation (TENS) in Children With Enuresis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 020891
Record Dates: First submitted 2015-11-03; First posted 2015-11-09 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2015-09

CONDITIONS: Enuresis; Nocturnal Enuresis; Urinary Incontinence
MeSH Terms: conditions — Enuresis; Nocturnal Enuresis; Urinary Incontinence | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TENS, 10 weeks (active) 2 hours a day. (Active Comparator): 26 children.
  Interventions: Device: Transcutaneous Electric Nerve Stimulation (TENS) - active
- TENS, 10 weeks (placebo) 2 hours a day. (Placebo Comparator): 26 children.
  Interventions: Device: Transcutaneous Electric Nerve Stimulation (TENS) - placebo

INTERVENTIONS:
Device: Transcutaneous Electric Nerve Stimulation (TENS) - active — TENS is a non-invasive method using surface electrodes. Except a few cases with local skin irritation in the area where the electrodes are applied, there is no evidence of side effects of TENS treatment.
  Arms: TENS, 10 weeks (active) 2 hours a day.
Device: Transcutaneous Electric Nerve Stimulation (TENS) - placebo
  Arms: TENS, 10 weeks (placebo) 2 hours a day.

SUMMARY:
This is a randomized, double blind, placebo controlled study of the effect of Sacral Transcutaneous Electric Nerve Stimulation (TENS) in fifty-two children with monosymptomatic nocturnal enuresis (MNE).

DETAILED DESCRIPTION:
Objectives:

Nighttime urinary incontinence (enuresis) is seen by 5-10% of children from six to fifteen years. Enuresis is a socially and psychologically stressful condition that can lead to bullying and low self esteem. Today the condition is treated with desmopressin or bells, that awake children at nighttime urination. One third of children suffering from enuresis are refractory to first line of treatment. Transcutaneous Electric Nerve Stimulation (TENS) has been documented efficacious on symptoms in children with daytime incontinence. Little is known regarding the effect of TENS on monosymptomatic nocturnal enuresis (MNE). The aim of our study is to investigate the effect of TENS on children diagnosed with MNE.

Methods:

This is a randomized, double blind, placebo controlled study of the effect of TENS in fifty-two children with MNE. The study period is from September 2015 to September 2016. The children recruited will receive TENS one hour during daytime and one hour during sleep for a total treatment period of ten weeks. The surface electrodes will be placed on the skin over s2-s3. TENS is safe and not associated with adverse effects.

Expected results:

The investigators hypothesize a reduction in number of wet nights in the enuretic children receiving active TENS. If TENS proves effective in children with enuresis it will be implemented as part of enuresis treatment in the clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Unremarkable clinical examination
* 3 or more wet nights per week
* No treatment of enuresis 1 week before the treatment starts (for bells two weeks)

Exclusion Criteria:

* Nighttime urine production on wet nights > 130 % of "maximum voided volume" (MVV) for age
* Ongoing constipation and/or faecal incontinence that are not successfully treated
* Daytime incontinence
* Prior or ongoing treatment with TENS
* Current or previous clinical history, clinical or laboratory findings or daily treatment with drugs that can be related to diseases or conditions that are expected to change the parameters investigated, especially diseases of the kidney and urinary tract or endocrine disorder
* Neurological and/or significant anatomical abnormalities of the urinary tract
* Previous operation in the urinary tract
* Recurrent urinary tract infections
* Incomplete bladder emptying (assessed with ultrasound) which means post micturition urine volume in the bladder > 20 ml or > 10 % of the total urine production

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2015-09; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Frequency of wet nights | 1 year
  Non-response is a reduction in wet nights < 50%, partial response a reduction of 50-89%, response a reduction of 90-99% and full response a reduction of 100% or less than one wet night in a month

SECONDARY OUTCOMES:
Maximum voided volume though daytime (MVV) | 1 year
Nighttime urine production (NUP) on wet nights | 1 year
Percent of wet night where NUP < MVV | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Søren Rittig, DMSc, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Skejby, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Publication

REFERENCES:
- [Background] Culbert TP, Banez GA. Wetting the bed: integrative approaches to nocturnal enuresis. Explore (NY). 2008 May-Jun;4(3):215-20. doi: 10.1016/j.explore.2008.02.014. No abstract available. PMID 18466855
- [Background] Hagglof B, Andren O, Bergstrom E, Marklund L, Wendelius M. Self-esteem in children with nocturnal enuresis and urinary incontinence: improvement of self-esteem after treatment. Eur Urol. 1998;33 Suppl 3:16-9. doi: 10.1159/000052236. PMID 9599731
- [Background] Kamperis K, Hagstroem S, Rittig S, Djurhuus JC. Combination of the enuresis alarm and desmopressin: second line treatment for nocturnal enuresis. J Urol. 2008 Mar;179(3):1128-31. doi: 10.1016/j.juro.2007.10.088. Epub 2008 Jan 18. PMID 18206924
- [Background] Yeung CK, Sreedhar B, Sihoe JD, Sit FK, Lau J. Differences in characteristics of nocturnal enuresis between children and adolescents: a critical appraisal from a large epidemiological study. BJU Int. 2006 May;97(5):1069-73. doi: 10.1111/j.1464-410X.2006.06074.x. PMID 16643494
- [Background] Rittig S, Frokiaer J. Basis and therapeutical rationale of the urinary concentrating mechanism. Int J Clin Pract Suppl. 2007 Sep;(155):2-7. doi: 10.1111/j.1742-1241.2007.01461.x. PMID 17727573
- [Background] Negoro H, Kanematsu A, Doi M, Suadicani SO, Matsuo M, Imamura M, Okinami T, Nishikawa N, Oura T, Matsui S, Seo K, Tainaka M, Urabe S, Kiyokage E, Todo T, Okamura H, Tabata Y, Ogawa O. Involvement of urinary bladder Connexin43 and the circadian clock in coordination of diurnal micturition rhythm. Nat Commun. 2012 May 1;3:809. doi: 10.1038/ncomms1812. PMID 22549838
- [Background] Bower WF, Moore KH, Adams RD, Shepherd R. A urodynamic study of surface neuromodulation versus sham in detrusor instability and sensory urgency. J Urol. 1998 Dec;160(6 Pt 1):2133-6. doi: 10.1097/00005392-199812010-00049. PMID 9817339
- [Background] Hasan ST, Robson WA, Pridie AK, Neal DE. Transcutaneous electrical nerve stimulation and temporary S3 neuromodulation in idiopathic detrusor instability. J Urol. 1996 Jun;155(6):2005-11. PMID 8618309
- [Background] Appell RA. Electrical stimulation for the treatment of urinary incontinence. Urology. 1998 Feb;51(2A Suppl):24-6. doi: 10.1016/s0090-4295(98)90004-8. PMID 9495731
- [Background] Hagstroem S, Mahler B, Madsen B, Djurhuus JC, Rittig S. Transcutaneous electrical nerve stimulation for refractory daytime urinary urge incontinence. J Urol. 2009 Oct;182(4 Suppl):2072-8. doi: 10.1016/j.juro.2009.05.101. Epub 2009 Aug 20. PMID 19695629
- [Background] Hagstroem S, Rittig N, Kamperis K, Mikkelsen MM, Rittig S, Djurhuus JC. Treatment outcome of day-time urinary incontinence in children. Scand J Urol Nephrol. 2008;42(6):528-33. doi: 10.1080/00365590802098367. PMID 18609267
- [Background] Bower WF, Moore KH, Adams RD. A pilot study of the home application of transcutaneous neuromodulation in children with urgency or urge incontinence. J Urol. 2001 Dec;166(6):2420-2. PMID 11696802
- [Background] Hoebeke P, Van Laecke E, Everaert K, Renson C, De Paepe H, Raes A, Vande Walle J. Transcutaneous neuromodulation for the urge syndrome in children: a pilot study. J Urol. 2001 Dec;166(6):2416-9. PMID 11696801
- [Background] De Gennaro M, Capitanucci ML, Mastracci P, Silveri M, Gatti C, Mosiello G. Percutaneous tibial nerve neuromodulation is well tolerated in children and effective for treating refractory vesical dysfunction. J Urol. 2004 May;171(5):1911-3. doi: 10.1097/01.ju.0000119961.58222.86. PMID 15076308
- [Background] Malm-Buatsi E, Nepple KG, Boyt MA, Austin JC, Cooper CS. Efficacy of transcutaneous electrical nerve stimulation in children with overactive bladder refractory to pharmacotherapy. Urology. 2007 Nov;70(5):980-3. doi: 10.1016/j.urology.2007.06.1109. Epub 2007 Oct 24. PMID 17919697
- [Background] Lordelo P, Teles A, Veiga ML, Correia LC, Barroso U Jr. Transcutaneous electrical nerve stimulation in children with overactive bladder: a randomized clinical trial. J Urol. 2010 Aug;184(2):683-9. doi: 10.1016/j.juro.2010.03.053. Epub 2010 Jun 18. PMID 20561643
- [Background] Lordelo P, Soares PV, Maciel I, Macedo A Jr, Barroso U Jr. Prospective study of transcutaneous parasacral electrical stimulation for overactive bladder in children: long-term results. J Urol. 2009 Dec;182(6):2900-4. doi: 10.1016/j.juro.2009.08.058. Epub 2009 Oct 28. PMID 19846164
- [Background] Tanagho EA, Schmidt RA. Electrical stimulation in the clinical management of the neurogenic bladder. J Urol. 1988 Dec;140(6):1331-9. doi: 10.1016/s0022-5347(17)42038-6. No abstract available. PMID 3057221
- [Background] Elabbady AA, Hassouna MM, Elhilali MM. Neural stimulation for chronic voiding dysfunctions. J Urol. 1994 Dec;152(6 Pt 1):2076-80. doi: 10.1016/s0022-5347(17)32312-1. PMID 7966678
- [Background] Bower WF, Yeung CK. A review of non-invasive electro neuromodulation as an intervention for non-neurogenic bladder dysfunction in children. Neurourol Urodyn. 2004;23(1):63-7. doi: 10.1002/nau.10171. PMID 14694460
- [Background] Neveus T, von Gontard A, Hoebeke P, Hjalmas K, Bauer S, Bower W, Jorgensen TM, Rittig S, Walle JV, Yeung CK, Djurhuus JC. The standardization of terminology of lower urinary tract function in children and adolescents: report from the Standardisation Committee of the International Children's Continence Society. J Urol. 2006 Jul;176(1):314-24. doi: 10.1016/S0022-5347(06)00305-3. PMID 16753432